CLINICAL TRIAL: NCT04001010
Title: Safety and Efficacy of PPP011-kit for Improving Physical Functioning and for Modulating Cachexia Progression in Patients With Advanced Cancer and Associated Cachexia: a Randomized, Double Blind, Placebo Controlled, Parallel Group Study
Brief Title: Safety and Efficacy of Inhaled Synthetic THC/CBD for Improving Physical Functioning and for Modulating Cachexia Progression in Patients With Advanced Cancer and Associated Cachexia
Acronym: SERENITY
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is postponed
Sponsor: Tetra Bio-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPP011-Ph3-01
Record Dates: First submitted 2019-05-31; First posted 2019-06-27 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Cannabis Use; Cachexia; Cancer; Advanced Cancer
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inhaled THC/CBD (PPP011) (Experimental): PPP011 (synthetic THC/CBD) inhalation with mighty medic device
  Interventions: Drug: PPP011
- Placebo (Placebo Comparator): Placebo inhalation with mighty medic device
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPP011 — 1 capsule inhaled 3 times a day with a vaporizer device
  Other Names: CAUMZ
  Arms: inhaled THC/CBD (PPP011)
Drug: Placebo — 1 capsule inhaled 3 times a day with a vaporizer device
  Arms: Placebo

SUMMARY:
A large number of patients with advanced cancer also suffer from cachexia. Cachexia is a syndrome characterized by loss of skeletal muscle mass (with/or without loss of fat mass) that cannot be reversed by nutritional support and progressively leads to functional impairment. Patients who suffer from anorexia and cachexia have lower survival rates. Some patients with cancer use cannabis to improve the way they feel and relieve their pain. However, there is very sparse high-quality research to prove that cannabis products are truly effective. This study will investigate patients with advanced cancer who use inhaled therapeutic cannabinoid-based medication (PPP011), in addition to palliative care management, and will assess if these patients experience improvement in functional status as a surrogate endpoint for survivalquality

DETAILED DESCRIPTION:
This is a 12-week randomized, double-blind, placebo-controlled, parallel group design trial to evaluate the safety and efficacy of inhaled PPP011 on physical functioning and cachexia progression in patients with cachexia related to advanced incurable cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent,
2. Adult male and female patients at least 18 years of age,
3. Patient agreed to follow the protocol,
4. Advanced cancer for which there is no known curative therapy,
5. The patient has a cachexia weight loss of Grade of 2 or Grade 3 cachexia as follow (based on Weight Loss Grading System) Weight loss accounts for the last 6 months before screening.
6. Patient's weight 6 months before screening must be available
7. Karnofsky Performance Status score ≥ 60 %
8. Life expectancy of at least 4 months, excluding refractory cachexia
9. No cognitive impairment according to Mini-Cog Negative confusion assessment according to CAM,
10. The patient is able to perform deep inhalations with FEV1 more than 60%,
11. Ability to read and respond to questions in French or English or French or Spanish,
12. A female volunteer must meet one of the following criteria:

If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose, If of non-childbearing potential - should be surgically sterile or in a menopausal state, A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must be surgically sterile or agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
physical functioning related to advanced cancer will be measured using a patient self rating questionnaire. | Change from baseline in EORTC-QLQ-C15-PAL physical functioning in multi-item scales at week 4, 8 and 12 W4 W8 W12
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 15 Palliative (EORTC-QLQ-C15-PAL). items are rated on a scale of 1 (not at all) to 4 (very much). high scores on a symptom scale correlate to increased symptom burden
Cachexia grade will be measured as per Weight Loss Grading System | Change from baseline at week 4, 8 and 12.
  Downgrading cachexia grade or grade maintenance will be considered as a drug benefit.

SECONDARY OUTCOMES:
pain will be recorded: VAS | Observed and Change from baseline in a VAS on pain AND no increase in pain medications at week 4, 8 and, 12 and 24.
  using a visual analogue scale. horizontal 0-100 mm VAS assessing pain
Patient nutritional and functional assessment will be meseared using a patient self rating questionnaire | Observed and change from baseline in patient nutritional and functional assessment (PG-SGA) at baseline and week 4, 8 and, 12.
  Patient-generated-subjective global assessment (PG-SGA) where critical need for nutrition intervention is defined as having a score ≥ 9 The higher the score the greater the risk for malnutrition

CONTACTS AND LOCATIONS:
Overall Officials: Martin Chasen, MD, Principal Investigator — William Osler Health Service Brampton
Locations (1):
- William Osler Health Service Brampton, Brampton, Ontario, Canada